CLINICAL TRIAL: NCT02685982
Title: Examining the Effects of Music and Rhythmic Sensory Stimulation on Major Depressive Disorder
Brief Title: Treating Major Depressive Disorder With Music and Low-frequency Rhythmic Sensory Stimulation
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University Health Network, Toronto (Other)
Collaborators: University of Toronto (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 15-9799
Record Dates: First submitted 2016-02-11; First posted 2016-02-19 (Estimated); Last update posted 2017-12-13 (Actual); Status verified 2016-10

CONDITIONS: Major Depressive Disorder
Keywords: Unipolar; Depression; Depressive Disorder; Behavioural Symptoms; Mood Disorder; Adjunctive Therapy; Music Therapy; Brain Stimulation
MeSH Terms: conditions — Depressive Disorder, Major; Depression; Depressive Disorder; Behavioral Symptoms; Mood Disorders

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Rhythmic Sensory Stimulation (Experimental): Participants in this group will undertake 30 minutes of daily Rhythmic Sensory Stimulation, for 5 day per week, for a total of 5 weeks. The stimulation consists of specially composed relaxing music tracks embedded with gamma frequency sounds of 30-70 Hz range. The intervention is conducted at the participant's home using a portable device called Sound Oasis Vibroacoustic Therapy System (VTS) 1000 unit. This device is a low-voltage consumer product device that has built in low frequency (subwoofer-type) speakers. The low frequency sounds played by the subwoofer speaker is experienced as vibrotactile vibration that is synchronized with the relaxing musical track.
  Interventions: Device: Rhythmic Sensory Stimulation

INTERVENTIONS:
Device: Rhythmic Sensory Stimulation — The stimulation consists of 30 minutes of daily stimulation with specially composed relaxing music tracks embedded with gamma frequency sounds of 30-70 Hz range.
  In this study, the stimuli will be delivered with a portable sound device called Sound Oasis Vibroacoustic Therapy System (VTS-1000) unit, which is a low-voltage consumer product that has two built in mid to high frequency speakers and one built in low frequency (subwoofer-type) speaker. The low frequency sounds played by the subwoofer speaker is experienced as vibrotactile vibration. Although the Intervention of Interest in this study is the Rhythmic Sensory Stimulation with low-frequency sounds, the efficacy of the Sound Oasis VTS-1000 device to deliver the intervention will also be subject to observation.

SUMMARY:
Major depressive disorder (MDD) is a highly prevalent and disabling disorder associated with persistent low mood, loss of the capacity to experience pleasure (i.e. anhedonia), reduced social functioning, and impaired quality of life. MDD is estimated to affect approximately 2% of Canadian women and 1% of Canadian men at any point in time. The World Health Organization affirms that depression is the leading cause of disability worldwide, with increasing global economic impact.

Standard treatments for depression include basic psychosocial support combined with antidepressant medication or psychotherapy. It has been observed, however, that only 50% of individuals respond to psychological treatment, and only 30-40% of patients achieve full remission after initial treatment with antidepressants. Music- and sound-related therapies have the potential to serve as adjuncts to, or facilitators of, medication.

In this study we will examine the effectiveness of a new therapeutic tool, known as Rhythmic Sensory Stimulation, as an adjunctive treatment for Major Depressive Disorder. Rhythmic Sensory Stimulation is a non-invasive brain stimulation technique that uses periodic pulses of light, sound, or tactile stimulus, to induce changes in the patterns of brain activity. Participants in this study will undertake 30 minutes of daily music intervention self-administered at home, for 5 days per week, for a total of 5 weeks. We will assess depression symptoms, sleep quality, quality of life, and brain activity pre- and post-treatment.

The results of the present study will help to better understand the effectiveness of Rhythmic Sensory Stimulation to the treatment of mood disorders, and contribute to the development of future studies to investigate the neural driving effects of therapies based on Rhythmic Sensory Stimulation.

DETAILED DESCRIPTION:
Major depressive disorder (MDD) is a highly prevalent and disabling disorder associated with persistent low mood, loss of the capacity to experience pleasure (i.e. anhedonia), reduced social functioning, and impaired quality of life. MDD is estimated to affect approximately 2% of Canadian women and 1% of Canadian men at any point in time. The World Health Organization affirms that depression is the leading cause of disability worldwide, with increasing global economic impact.

Standard treatments for depression include basic psychosocial support combined with antidepressant medication or psychotherapy. It has been observed, however, that only 50% of individuals respond to psychological treatment, and only 30-40% of patients achieve full remission after initial treatment with antidepressants. Music- and sound-related therapies have the potential to serve as adjuncts to, or facilitators of, medication. Several recent systematic reviews have concluded that music is an effective therapeutic tool with significant results on improving global state, symptoms, and overall functioning, and is also well-accepted by patients.

The goal of this project is to evaluate the effectiveness of music and rhythmic sensory stimulation with low-frequency sounds as an adjunctive therapy for depression. Through a systematic collection of clinical, behavioural and electrophysiological measures, the project also aims to determine the possible mechanisms that underlie the effects of music- and sound-based therapies on symptoms of MDD. In addition to measures of depression severity and symptoms, we are also interested in secondary behavioral measures addressing possible confounding variables, such as anhedonia, quality of life, and individual differences in how people experience reward and pleasure associated with music. These assessments will allow an initial investigation of the neural correlates of the therapeutic effects of music in the treatment of depression, which is greatly warranted to better understand the efficacy of music- and sound-based treatments.

ELIGIBILITY:
Inclusion Criteria:

* Outpatients 18 to 60 years of age.
* Meet DSM-IV-TR criteria for major depressive episode (MDE) in major depressive disorder (MDD) without psychotic features, as determined by clinician assessment.
* Episode duration > 3 months.
* MADRS score ≥ 15 (mild to severe symptoms intensity).
* Fluency in English, sufficient to complete the interviews and self-report questionnaires.
* Satisfactory hearing bilaterally based on self-report.

Exclusion Criteria:

* Any Axis I diagnosis (other than MDD), and MDD with psychotic features,that is considered the primary diagnosis.
* Fibromyalgia diagnosis (FIQR score ≥ 39).
* Bipolar-I or Bipolar-II diagnosis (HCL score ≥ 14).
* Presence of a significant Axis II diagnosis (borderline, antisocial), judged as being primary based on clinician assessment.
* High suicidal risk, defined by clinician judgment.
* Substance dependence/abuse in the past 6 months.
* Presence of significant neurological disorders, head trauma, or other unstable medical conditions.
* Acute and active inflammatory conditions, rheumatoid arthritis, osteoarthritis, autoimmune disease.
* History of epilepsy, seizures.
* Hemorrhaging or active bleeding.
* Hearing impairment.
* Thrombosis or heart diseases, including hypotension, arrhythmia, pacemaker, angina pectoris.
* Pregnant or breastfeeding.
* Recovering from recent accident with prolapsed vertebral disc, back or neck injury.
* Started psychological treatment within the past 3 months with the intent of continuing treatment.
* Patients who have changed medication or adjusted medication dosage within 4 weeks.

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 20 (Actual)
Dates: Start 2016-04 (Actual); Primary Completion 2017-08 (Actual); Study Completion 2017-08 (Actual)

PRIMARY OUTCOMES:
Change in MADRS (Montgomery-Asberg Depression Rating Scale) scores from baseline | Assessed at Week 0 (pre-intervention) and Week 6 (post-intervention)
  Clinical response (≥ 50% reduction in MADRS scores from baseline)

CONTACTS AND LOCATIONS:
Overall Officials: Sidney H Kennedy, MD, Principal Investigator — University Health Network, Toronto; Lee Bartel, PhD, Principal Investigator — University of Toronto

IPD SHARING:
Plan to Share IPD: Yes
Data will be stored and shared through Ontario Brain Institute platform (BRAIN-Code).